CLINICAL TRIAL: NCT00180401
Title: MODULA-Study: Modul 10: Benefit of CRT-therapy in CRT-Patients With QRS-complex of 120 - 150 ms
Status: Terminated | Type: Observational
Why Stopped: no longer interest from medical community
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Guidant Corporation (Industry)
Other Study IDs: Version vom 05.08.2002
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- QRS 120-150 ms: Subjects with a QRS width between 120-150 ms
  Interventions: Behavioral: CRT-P and CRT-D devices
- QRS >150 ms: Subjects with a QRS width >150 ms
  Interventions: Behavioral: CRT-P and CRT-D devices

INTERVENTIONS:
Behavioral: CRT-P and CRT-D devices

SUMMARY:
The purpose of this study is to compare the benefit of cardiac resynchronization therapy (CRT)-therapy in patients with a QRS-complex of 120-150 ms to patients with a QRS-complex of > 150 ms.

DETAILED DESCRIPTION:
The objective of this study is to compare the benefit of CRT-therapy in patients with a QRS-complex of 120-150 ms to patients with a QRS-complex of > 150 ms within 12 months. A benefit is defined as change in quality of life and change in physical ability.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiac resynchronization therapy with a defibrillator (CRT-D) or cardiac resynchronization therapy pacemakers (CRT-P) system
* New York Heart Association (NYHA) III
* Ejection fraction (EF) below 35%
* Optimised medical therapy
* QRS-complex above 120 ms

Exclusion Criteria:

* Patients with CRT-P and atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-06; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Observational: Benefit of CRT | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Tiroke, MD, Principal Investigator — Klinikum der Christian Albrecht Universität / Kardiologische Abteilung / Arnold Heller-Str. 7 / 24105 Kiel / Germany
Locations (1):
- Klinikum der Christian Albrecht Universität / Kardiologische Abteilung, Kiel, Germany